CLINICAL TRIAL: NCT00842257
Title: A Single Arm Phase II Trial of Panitumumab in Cetuximab Refractory KRAS Wild-Type Colorectal Cancer
Brief Title: Panitumumab in Cetuximab Refractory KRAS Wild-Type Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Dana-Farber Cancer Institute (Other); Amgen (Industry)
Responsible Party: Principal Investigator, David Patrick Ryan, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-287; 20070602 (Other: Amgen)
Record Dates: First submitted 2009-02-10; First posted 2009-02-12 (Estimated); Results first posted 2017-05-16 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-04

CONDITIONS: Colorectal Cancer
Keywords: panitumumab; cetuximab; KRAS wild-type
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Panitumumab (Experimental): Panitumumab administered by a central line infusion on days 1 and 15 of each 4 week cycle.
  Interventions: Drug: panitumumab

INTERVENTIONS:
Drug: panitumumab — Panitumumab is administered intravenously (IV) by an infusion pump through a peripheral line or indwelling catheter using a 0.2 or 0.22-micron in-line filter infusion set-up over 1 hour 15 minutes. The starting panitumumab dose is 6 mg/kg administered every 14 days for as long as patients are on study without evidence of disease progression or demonstrating intolerance to treatment. The total dose may be rounded up or down by no greater than 10 mg. The panitumumab dose will be calculated based on the subject's actual body weight at each visit. Panitumumab will be diluted in a minimum of 100 mL of pyrogen-free 0.9% sodium chloride solution (normal saline solution, supplied by the site). The maximum concentration of the diluted solution to be infused should not exceed 10 mg/mL.
  Other Names: Vectibix

SUMMARY:
The purpose of this research study is to learn whether panitumumab helps treat colorectal cancer in participants who have not responded to treatment with cetuximab. Panitumumab is a human monoclonal antibody. Antibodies are proteins that recognize a foreign substance in the body and then attach themselves to it making it exposed to destruction. Panitumumab attaches itself to a protein on cancer cells called "epidermal growth factor receptor" or EGFR. EGFR helps cancer cells to grow, and blocking EGFR helps prevent cancer cells from growing.

DETAILED DESCRIPTION:
* Panitumumab will be given to the participants through a central line. A central line is a long, thin tube (catheter) that is inserted through the skin into a large vein in the chest. This is placed by a radiologist or surgeon.
* Panitumumab will be given in 4-week cycles. Panitumumab infusions will be given on days 1 and 15 of each cycle (every 2 weeks).
* The following procedures will be performed on days 1 and 15 of each cycle, before each infusion: physical exam; questions about any symptoms or side effects; performance status; routine blood tests and CT or MRI (every 2 cycles).
* Participants can continue to receive panitumumab until their disease gets worse or they experience unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of colorectal adenocarcinoma and measurable disease by RECIST criteria on CT or MRI
* Treated with cetuximab as part of their last treatment regimen for at least 4 weeks and must have been taken off cetuximab therapy for disease progression. Patients may or may not have been treated with 5-FU (5-Fluorouracil), oxaliplatin, irinotecan and bevacizumab. There is no maximal number of pre-existing treatment regimens. At least 2 weeks must have elapsed between previous anticancer therapy and the start of treatment on protocol, AND resolution of any skin rash related to prior treatment with epidermal growth factor receptor inhibitor
* ECOG (Eastern Cooperative Oncology Group) Performance Status 0, 1 or 2
* Life expectancy of greater than 3 months
* Normal organ, metabolic, and marrow function as defined in the protocol
* A wild-type tumor K-RAS gene (Kirsten rat sarcoma viral oncogene homolog) as determined by sanger sequencing of exon 2 from tumor DNA
* 18 years of age or older

Exclusion Criteria:

* History of untreated and or progression central nervous system metastases
* History of another primary cancer except: curatively treated in situ cervical cancer or breast; curatively resected non-melanoma skin cancer; other primary solid tumor curatively treated with no known active disease present and no treatment administered for 3 years or more prior to enrollment
* Intolerance to cetuximab leading to drug discontinuation due to rash, GI toxicity, or other grade 3 or 4 toxicities
* Radiotherapy < 14 days prior to enrollment
* Systemic chemotherapy, hormonal therapy, immunotherapy, or experimental or approved proteins/antibodies < 14 days before enrollment
* Subjects requiring chronic use of immunosuppressive agents
* Any investigational agent or therapy 30 days prior to enrollment
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with any study requirements
* History of interstitial lung disease
* Women who test positive for serum or urine pregnancy test or who are breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-05 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aram Hezel, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wadlow RC, Hezel AF, Abrams TA, Blaszkowsky LS, Fuchs CS, Kulke MH, Kwak EL, Meyerhardt JA, Ryan DP, Szymonifka J, Wolpin BM, Zhu AX, Clark JW. Panitumumab in patients with KRAS wild-type colorectal cancer after progression on cetuximab. Oncologist. 2012;17(1):14. doi: 10.1634/theoncologist.2011-0452. Epub 2011 Dec 30. PMID 22210091

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects identified by their treating oncologist in the Gastrointestinal Cancer Clinics at Massachusetts General Hospital and Dana-Farber Cancer Institute, all therapy options are discussed (including participation in this trial).
Groups:
- Panitumumab: Panitumumab administered by a central line infusion over 1 hour 15 minutes on days 1 and 15 of each 4 week cycle. The starting panitumumab dose is 6 mg/kg, the total dose may be rounded up or down by no greater than 10 mg. The panitumumab dose is calculated based on the subject's actual body weight at each visit. Panitumumab is diluted in a minimum of 100 mL of pyrogen-free 0.9% sodium chloride solution. The maximum concentration of the diluted solution to be infused should not exceed 10 mg/mL.
Period: Overall Study
Arm/Group | Panitumumab
Started | 20
Completed | 19
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Panitumumab
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 54.5 [39 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20
ECOG PS [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group Performance Status. 0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  Participants
    0 | 4
    1 | 14
    2 | 2
Primary tumor [Count of Participants; unit: Participants]
  Colon | 17
  Rectal | 3
Metastatic sites [Number; unit: participants]
  Liver | 15
  Lung | 11
  Lymph Nodes | 9
Prior therapy [Number; unit: participants]
  Cetuximab | 20
  Flouropyrimidine | 20
  Oxaliplatin | 19
  Irinotecan | 18
  Bevacizumab | 17

OUTCOME MEASURES:

1. Primary Outcome: Response Rate of Single Agent Panitumumab Among Patients With KRAS Wild-type Colorectal Cancer Previously Treated With Cetuximab.
Description: The response rate of single agent panitumumab among patients with KRAS wild-type (Kirsten rat sarcoma viral oncogene homolog) colorectal cancer previously treated with cetuximab. Inclusive of three patients with clinical progression prior to first re-staging CT scans. Response rate evaluated using RECIST (Response Evaluation Criteria In Solid Tumors). Best overall response is recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
  RECIST:
  Complete Response (CR): Disappearance of all target lesions Partial Response (PR): At least a 30% decrease in the sum of the LD (longest diameter) of target lesions Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions
Time Frame: 3 years
Population: One patient withdrawn for an infusion reaction prior to first re-staging CT scans.
Measure: Count of Participants; unit: Participants
Arm/Group | Panitumumab
Number analyzed (Participants) | 19
Participants
  Partial Response | 0
  Stable Disease | 9
  Progressive Disease | 10

2. Secondary Outcome: Median Progression Free Survival (PFS)
Description: The duration of time from start of treatment to time of radiologic disease progression per RECIST or death, or otherwise the date of last tumor assessment. Median PFS was calculated using Kaplan Meier suvival analysis. Progressive disease is defined as having at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: 3 years
Population: One patient withdrawn due to an infusion reaction prior to first re-staging CT scans.
Measure: Median (Full Range); unit: Months
Arm/Group | Panitumumab
Number analyzed (Participants) | 19
Months | 1.7 [0.5 to 3.7]

3. Secondary Outcome: Median Overall Survival
Description: The duration of time from start of treatment to time of death or otherwise the date of last tumor assessment. Median survival was calculated using Kaplan Meier suvival analysis.
Time Frame: 3 years
Measure: Median (Full Range); unit: Months
Arm/Group | Panitumumab
Number analyzed (Participants) | 20
Months | 5.2 [1 to 18.2]

4. Secondary Outcome: Disease Control Rate as Defined by RECIST Criteria
Description: Disease Control Rate as defined by RECIST criteria. The number patients achieving stable disease, partial response, or complete response at some point during follow-up.
Time Frame: 3 years
Population: One patient withdrawn for an infusion reaction prior to first re-staging CT scans.
Measure: Count of Participants; unit: Participants
Arm/Group | Panitumumab
Number analyzed (Participants) | 19
Participants | 9

ADVERSE EVENTS:
Time Frame: 3 Years
Description: Participants were assessed for toxicity before each dose.
Arm/Group | Panitumumab
All-Cause Mortality (participants affected / at risk) | 20/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 20/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panitumumab (N=20)
Abdomen- pain (Gastrointestinal disorders) | 5 (6)
Alkaline phosphatase (Metabolism and nutrition disorders) | 6 (11)
Allergic reaction (Immune system disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (4)
Anorexia (Gastrointestinal disorders) | 6 (7)
AST- SGOT (Metabolism and nutrition disorders) | 5 (8)
Back- pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bicarbonate (Metabolism and nutrition disorders) | 3 (4)
Bilirubin (Metabolism and nutrition disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 8 (8)
Creatinine (Metabolism and nutrition disorders) | 3 (5)
Dehydration (Gastrointestinal disorders) | 2 (2)
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 3 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (11)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Edema limb (Blood and lymphatic system disorders) | 3 (5)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 (5)
Fatigue (General disorders) | 15 (22)
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 2 (4)
Hemoglobin (Blood and lymphatic system disorders) | 7 (8)
Hemoglobinuria (Metabolism and nutrition disorders) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (7)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (7)
Hypermagnesemia (Metabolism and nutrition disorders) | 5 (5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (8)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 8 (15)
Hypophosphatemia (Metabolism and nutrition disorders) | 8 (13)
Insomnia (General disorders) | 4 (4)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2)
Neuropathy-sensory (Nervous system disorders) | 5 (5)
Pain-other (General disorders) | 3 (3)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4 (7)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 8 (18)
Weight loss (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No